CLINICAL TRIAL: NCT04716842
Title: Evaluation of Plasma Angiotensin II and Angiotensin II Receptor Levels in Patients With Sepsis and Septic Shock: a Prospective Observational Study.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ayse Belin Ozer, Prof. Dr., Inonu University
Other Study IDs: AOzer2
Record Dates: First submitted 2021-01-16; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Sepsis; Septic Shock
Keywords: sepsis; septic shock; angiotensin II
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- sepsis: In intensive care patients with suspected or proven infection, if the SOFA score ≥2, the patients will be evaluated as sepsis and routine examination, monitoring and treatment will be applied.
- septic shock: Patients with sepsis who require vasopressor to keep mean arterial pressure above 65 mmHg and lactate> 2 mmol/l will be included in the septic shock group.
- control: It will be formed from patients who are hospitalized in the intensive care unit for a reason other than sepsis and septic shock, without suspected or proven infection.

SUMMARY:
Evaluation of plasma angiotensin II and angiotensin II receptor levels in patients with sepsis and septic shock: a prospective observational study.

DETAILED DESCRIPTION:
There is an increasing number of experimental publications investigated effects of angiotensin II and receptors on the pathogenesis and treatment of sepsis and septic shock. However, its level in humans and its relationship with the severity of the disease has not been investigated. If angiotensin II plays a role in the diagnosis and prognosis of septic shock by evaluating this relationship in our study, it may be a biomarker to be used in future diagnosis, prediction of prognosis and treatment. This will enable early recognition and treatment of this disease, which causes high mortality and cost in intensive care units, thus increasing the survival rate and reducing the cost.

ELIGIBILITY:
Inclusion Criteria:

* intensive care unit patient

Exclusion Criteria:

* End-stage organ failure,
* immunodeficiency, vasospastic disease, pregnancy, other shock causes (hypovolemic, cardiogenic, neurogenic) a life expectancy of less than 48 hours

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Group sepsis (n = 25): In intensive care patients with suspected or proven infection, if the SOFA score ≥2, the patients will be evaluated as sepsis and routine examination, monitoring and treatment will be applied.
  Group septic shock (n = 25): Patients with sepsis who require vasopressor to keep mean arterial pressure above 65 mmHg and lactate> 2 mmol/l will be included in the septic shock group.
  Group Control (n = 25): It will be formed from patients who are hospitalized in the intensive care unit for a reason other than sepsis and septic shock, without suspected or proven infection.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
angiotensin II levels | 0-3 days
  serum angiotensin II levels
angiotensin II receptor I | 0-3 days
  serum angiotensin II receptor I levels
angiotensin II receptor II | 0-3 days
  serum angiotensin II receptor II levels

SECONDARY OUTCOMES:
procalsitonine level | 0-3 days
  Procalsitonine level
crp level | 0-3 days
  crp levels
mortality | 28 days
  mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Belin B OZER, Principal Investigator — Inonu University Faculty of Medicine
Locations (1):
- Ayse Belin B OZER, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided